CLINICAL TRIAL: NCT06067295
Title: Longitudinal Advanced Prostate Cancer Cohort (LAPCC)
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4P-22-2; NCI-2023-01434 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-22-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood and urine sample collection, complete surveys, and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study examines information from patients with prostate cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). By collecting biological samples (like blood, urine, and tissue), and health information (such as treatment, diet, and quality of life) researchers hope to learn more about prostate cancer and ways to improve outcomes in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To create an annotated biorepository with prospectively collected blood and urine samples from men with advanced prostate cancer.

OUTLINE: This is an observational study.

Patients undergo blood and urine sample collection, complete surveys, and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Men of all racial and ethnic groups 18 years of age or older
* Men with a diagnosis of advanced (metastatic) prostate cancer who are scheduled to begin a new systemic treatment (including first or subsequent lines of therapy)
* Prior participation on clinical trials is allowed

Exclusion Criteria:

* Inability to give informed consent
* Any other malignancy, unless previously treated with curative intent and the subject has been disease free for 3 years or longer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men diagnosed with advanced (metastatic) prostate cancer at Norris Comprehensive Cancer Center and Los Angeles General Medical Center with either metastatic castrate sensitive prostate cancer (mCSPC) or metastatic castration-resistant prostate cancer (mCRPC).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2027-02-21 (Estimated)

PRIMARY OUTCOMES:
Collection of biological specimens and clinical data for future research related to prostate cancer. | Up to 5 years
  The objective of this study is to create a biorepository of biospecimen and clinical data. There is no primary clinical outcome for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goldkorn, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California